CLINICAL TRIAL: NCT00455546
Title: PLASMA Trial: Phospholipase Levels And Serological Markers of Atherosclerosis: A Dose-Response Clinical Pharmacology Study of A-002 In Subjects With Stable Coronary Artery Disease
Brief Title: PLASMA Trial: A Dose-Response Study of A-002 In Subjects With Stable Coronary Artery Disease
Acronym: PLASMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-CVD-2221
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary; Artery; Atherosclerosis; Phospholipase; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — varespladib methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: A-002

SUMMARY:
The study will be conducted at up to 80 centers worldwide and will be a double-blind randomized parallel group placebo controlled study among subjects with stable coronary artery disease (CAD). Subjects will be randomized to receive either placebo tablets or one of 4 orally active doses of A-002. The duration of study drug therapy will be 8 weeks.

DETAILED DESCRIPTION:
A-002 represents a novel therapy for the treatment of atherosclerosis and coronary artery disease (CAD). Through the inhibition of activity A-002 may provide multifunctional activity directed against key facets of the disease process, namely a) inflammation, b) atherogenic lipid profiles and c) the atherosclerotic process. Non-clinical and clinical data from recent studies have demonstrated the benefit of early and aggressive anti-inflammatory therapy to reduce cardiovascular risk. Recent clinical studies have provided a strong association between levels and cardiovascular event risk. The proposed Phase 2 clinical pharmacology study (Study No. AN-CVD-2221) will examine the effects of 4 different doses of A-002 compared with placebo, on enzyme levels and activity after 8 weeks of treatment. In addition, the effect of treatment on inflammatory markers of cardiovascular risk (C-reactive protein [CRP]), lipid levels and lipoprotein subclasses and other soluble biomarkers (e.g., ICAM-1, VCAM-1, TNF, MCP-1 etc) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion if they meet the following inclusion criteria:

* Men and women > 18 years of age
* Written informed consent from the subject
* Stable CAD
* Stable medical condition, will be compliant and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subjects must NOT meet any of the following exclusion criteria:
* Planned CABG
* Hospitalization for acute coronary syndrome if troponin level is >0.1 ng/mL in the preceding 6 weeks
* Hospitalization for ST-segment acute myocardial infarction (STEMI) in the preceding 12 weeks
* Subjects with chronic inflammatory disease (e.g., RA), inflammatory bowel disease, recent (12 weeks) systemic or localized infection (the latter requiring clinical intervention), or major surgery
* hs-CRP >15 mg/L repeated on at least 2 occasions >24 hours apart due to non-cardiovascular systemic inflammatory conditions (e.g., rheumatoid disease)
* Acute or chronic heart failure as defined by the NYHA classification as functional Class III or Class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-04; Study Completion 2007-09

PRIMARY OUTCOMES:
Comparison of active and placebo treatments with respect to change from Baseline to Week 8 in sPLA2 levels and activity.

SECONDARY OUTCOMES:
Comparison of active and placebo treatments with respect to change in: Inflammatory markers, lipid and biochemical parameters, and LDL and HDL subclasses.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (23):
  - Mobile Heart Specialists, Mobile, Alabama
  - Sonoran Health Specialists, Scottsdale, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Hudson, Florida
  - Charlotte Cardiovascuar Research, Port Charlotte, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Augusta Cardiology Clinic, PC, Augusta, Georgia
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Cardiology, PC, Syracuse, New York
  - Oklahoma Cardiovascular and Hypertension Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Camp Hill, Pennsylvania
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - Austin Heart, Austin, Texas
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Winsconin Heart, SC, Madison, Wisconsin
- Ukraine (13):
  - Strazhesko Institute of Cardiology AMS, Kyiv, 03680
  - Dnipropetrovs'k State Medical Academy, Dnepropetrovs'k
  - Institute of Therapy of AMS, Kharkiv
  - Central Clinical Hospital "Ukrzaliznysti", Khirkov
  - Strazhesko Institute of Cardiology AMS, Kviv
  - Kiev Central Hospital #1, Kyiv
  - City Clinical Hospital No 12, Kyiv
  - Scientific Centre of Endocrine Surgery, Kyiv
  - Strazhesko Institute of Cardiology AMS, Kyiv
  - Institute of Gerontology AMS, Kyiv
  - Institute of Gerontology, Kyiv
  - L'viv Regional State Clinical Treatment and Diagnostics, Lviv
  - Hospital of "Radioprylad" Plant, Zaporizhzhya

REFERENCES:
- [Derived] Rosenson RS, Hislop C, McConnell D, Elliott M, Stasiv Y, Wang N, Waters DD; PLASMA Investigators. Effects of 1-H-indole-3-glyoxamide (A-002) on concentration of secretory phospholipase A2 (PLASMA study): a phase II double-blind, randomised, placebo-controlled trial. Lancet. 2009 Feb 21;373(9664):649-58. doi: 10.1016/S0140-6736(09)60403-7. PMID 19231633